CLINICAL TRIAL: NCT06553105
Title: Department of Radiology, School of Medicine, 5th Azar Hospital, Gorgan, Golestan, Iran
Brief Title: Diagnosis and Clinical Presentation of Iliac Graft-Enteric Fistula: A Case Report
Status: Not yet recruiting | Type: Observational
Sponsor: Golestan University of Medical sciences (Other)
Responsible Party: Principal Investigator, Reza zahedpasha, Department of Radiology, School of Medicine, 5th Azar Hospital, Gorgan, Golestan, Iran, Golestan University of Medical sciences
Other Study IDs: there is no id
Record Dates: First submitted 2024-08-10; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Case-report; Diagnosis; Digestive System Fistula; Gastrointestinal Hemorrhage; Iliac Graft-Enteric Fistula
Keywords: case-report; CT scan; Diagnosis; Digestive System Fistula; Gastrointestinal Hemorrhage; Iliac Graft-Enteric Fistula.
MeSH Terms: conditions — Disease; Digestive System Fistula; Gastrointestinal Hemorrhage | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ct scan — use ct scan for diagnosis fistula

SUMMARY:
Abstract

Introduction:

Aorto-enteric fistula (AEF) is a life-threatening complication arising from abnormal connections between the gastrointestinal tract and major arteries. One uncommon type, iliac artery-enteric fistula (IEF), can occur following vascular interventions such as arterial stent-graft placement.

Case Presentation:

We report the case of a 47-year-old male presenting with hematemesis and abdominal pain, who was diagnosed with an iliac graft-enteric fistula. Timely recognition and management were crucial for a favorable outcome.

Clinical Discussion:

Diagnosing AEFs remains challenging, requiring a multidisciplinary approach and high clinical suspicion. While computed tomography angiography (CTA) is commonly used for diagnosis, its sensitivity may be limited, emphasizing the importance of integrating clinical history and findings. Management strategies vary based on etiology and patient status, with surgery being pivotal.

Conclusion:

Aorto-enteric fistula, which can arise from a thrombosed graft, presents diagnostic challenges due to its rare formation. In patients with a history of vascular interventions and gastrointestinal bleeding, AEF should be considered. This case underscores the need for heightened awareness among healthcare professionals regarding AEF diagnosis and management to reduce severe morbidity, mortality, and prolonged hospital stays.

ELIGIBILITY:
Inclusion Criteria:

n/a

Exclusion Criteria:

n/a

Ages: 40 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: one man
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2024-08-11 (Estimated); Primary Completion 2024-08-12 (Estimated); Study Completion 2024-08-13 (Estimated)

PRIMARY OUTCOMES:
diagnosis of fistula by ct scan | one day